CLINICAL TRIAL: NCT03548090
Title: The Effects of Plantar Flexion Training on Plantar Flexion Activation, Torque, and Step Length Asymmetry in People With Chronic Stroke
Brief Title: The Effects of Plantar Flexion Training in People With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Daniel Wingard, Physical therapist, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MH-17-0284
Record Dates: First submitted 2018-05-24; First posted 2018-06-07 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Stroke; Hemiplegic Gait
Keywords: stroke rehabilitation; walking limitations; gait rehabilitation
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic | interventions — Weights and Measures; Clinical Trials, Phase I as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (24):
- 1 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 0 degrees, then 5 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 50%, then 75%, then 90%), Phase 3 (control 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Control 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 2 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 0 degrees, then 5 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 50%, then 90%, then 75%), Phase 3 (control 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Control 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 3 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 0 degrees, then 5 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 75%, then 50%, then 90%), Phase 3 (control 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Control 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 4 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 0 degrees, then 5 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 75%, then 90%, then 50%), Phase 3 (control 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Control 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 5 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 0 degrees, then 5 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 90%, then 50%, then 75%), Phase 3 (control 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Control 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 6 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 0 degrees, then 5 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 90%, then 75%, then 50%), Phase 3 (control 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Control 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 7 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 5 degrees, then 0 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 50%, then 75%, then 90%), Phase 3 (control 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Control 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 8 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 5 degrees, then 0 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 50%, then 90%, then 75%), Phase 3 (control 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Control 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 9 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 5 degrees, then 0 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 75%, then 50%, then 90%), Phase 3 (control 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Control 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 10 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 5 degrees, then 0 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 75%, then 90%, then 50%), Phase 3 (control 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Control 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 11 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 5 degrees, then 0 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 90%, then 50%, then 75%), Phase 3 (control 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Control 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 12 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 5 degrees, then 0 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 90%, then 75%, then 50%), Phase 3 (control 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Control 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 13 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 0 degrees, then 5 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 50%, then 75%, then 90%), Phase 3 (experimental 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Experimental 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 14 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 0 degrees, then 5 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 50%, then 90%, then 75%), Phase 3 (experimental 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Experimental 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 15 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 0 degrees, then 5 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 75%, then 50%, then 90%), Phase 3 (experimental 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Experimental 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 16 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 0 degrees, then 5 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 75%, then 90%, then 50%), Phase 3 (experimental 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Experimental 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 17 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 0 degrees, then 5 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 90%, then 50%, then 75%), Phase 3 (experimental 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Experimental 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 18 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 0 degrees, then 5 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 90%, then 75%, then 50%), Phase 3 (experimental 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Experimental 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 19 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 5 degrees, then 0 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 50%, then 75%, then 90%), Phase 3 (experimental 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Experimental 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 20 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 5 degrees, then 0 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 50%, then 90%, then 75%), Phase 3 (experimental 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Experimental 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 21 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 5 degrees, then 0 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 75%, then 50%, then 90%), Phase 3 (experimental 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Experimental 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 22 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 5 degrees, then 0 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 75%, then 90%, then 50%), Phase 3 (experimental 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Experimental 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 23 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 5 degrees, then 0 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 90%, then 50%, then 75%), Phase 3 (experimental 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Experimental 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise
- 24 (Experimental): Phase 1 (skateboard exercise at 50% body weight and an incline level of 5 degrees, then 0 degrees), Phase 2 (skateboard exercise with incline level determined to be optimal in phase 1 and body weight at 90%, then 75%, then 50%), Phase 3 (experimental 4-week exercise intervention)
  Interventions: Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight; Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight; Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight; Other: Experimental 4-week exercise intervention; Other: Over-ground multi-directional gait training; Other: Home exercise

INTERVENTIONS:
Other: Skateboard exercise at an incline angle of 0 degrees and 50% body weight — Participants will stand on a specified incline angle (0 degrees) and with a specified body weight (50%) on the paretic LE and will simultaneously move a small skateboard forward with the non-paretic LE.
Other: Skateboard exercise at an incline angle of 5 degrees and 50% body weight — Participants will stand on a specified incline angle (5 degrees) and with a specified body weight (50%) on the paretic LE and will simultaneously move a small skateboard forward with the non-paretic LE.
Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 75% body weight — Participants will stand on a specified incline angle (either 0 or 5 degrees, whichever is determined during phase 1 to be optimal) and with a specified body weight (75%) on the paretic LE and will simultaneously move a small skateboard forward with the non-paretic LE.
Other: Skateboard exercise at an incline angle determined to be optimal in phase 1 (either 0 or 5 degrees) and 90% body weight — Participants will stand on a specified incline angle (either 0 or 5 degrees, whichever is determined during phase 1 to be optimal) and with a specified body weight (90%) on the paretic LE and will simultaneously move a small skateboard forward with the non-paretic LE.
Other: Control 4-week exercise intervention — This intervention occurs in phase 3. Subjects will participate in 1-hour sessions three times per week for four weeks. The control group will perform three sets of ten repetitions of the following 4 exercises, for a total of 120 repetitions: 1) standing hip abduction against green theraband resistance with upper extremity support, 2) sit to stands from chair with no upper extremity support, 3) bilateral calf raises with upper extremity support, and 4) right and left weight shifting exercises using a wobble board with upper extremity support available if needed.
  Other Names: conventional physical therapy
  Arms: 1; 10; 11; 12; 2; 3; 4; 5; 6; 7; 8; 9
Other: Experimental 4-week exercise intervention — This intervention occurs in phase 3. Subjects will participate in 1-hour sessions three times per week for four weeks. The experimental group will perform the skateboard exercise with the optimal parameters established during studies 1 and 2 (that is, an incline angle of either 0 or 5 degrees and a body weight percentage of 50%, 75%, or 90%)--the forward and backward speed of the skateboard will be cued with a metronome that will set at a beats per minute that matches the foot strike cadence of someone walking at 0.7 m/s, and the magnitude of forward excursion of the skateboard will be individualized to the participant based on GAITRite® data (that is, step length of the non-paretic LE).
  Other Names: Plantar flexion training
  Arms: 13; 14; 15; 16; 17; 18; 19; 20; 21; 22; 23; 24
Other: Over-ground multi-directional gait training — In the over-ground multi-directional gait protocol, the participant will walk 750 steps forward, 50 steps backward, and 200 side steps over level surfaces. The over ground gait training will focus on equalizing step length while performing multi-directional gait training.
Other: Home exercise — Home exercise consists of three sets of ten repetitions of the following three exercises to be performed on non-therapy days over the four weeks of phase 3: 1) sit to stands from chair with no upper extremity support, 2) bilateral calf raises with hand support, and 3) resisted side stepping to the non-paretic side using a green theraband with upper extremity support.

SUMMARY:
This study consists of three phases that aim to develop an exercise intervention to promote maximal activation of ankle plantar flexors in the paretic lower extrimty (LE) in order to restore a more normalized gait pattern in chronic stroke survivors.

The aim of the first phase is to determine if there are differences between standing on different levels of inclination on plantar flexion activation during forward movement of the contralateral LE in adults with chronic with stroke.

The aim of second phase is to determine if there are differences between different percentages of weight bearing on the paretic LE on plantar flexion activation during forward movement of the contralateral LE in adults with chronic stroke.

The aim of the third phase is to determine if there are differences between a 4-week plantar flexion training intervention and conventional physical therapy.

DETAILED DESCRIPTION:
Description of Arms:

This study has three phases. The first phase is performed in a cross-over fashion. Participants will stand on two different incline angles on the paretic LE and simultaneously move a small skateboard forward with the non-paretic LE. The testing order for the two different incline angles will be randomized, and all participants will be required to complete both incline angle conditions within a single test session.

The second phase will also be performed in a cross-over fashion. Participants will stand with three different percentages of body weight on their paretic LE while moving the skateboard forward with the non-paretic LE. The testing order for the three body weight percentages will be randomized. All participants will be required to complete all three body weight conditions within a single test session.

In the third phase, participants will be randomized to either a control 4-week exercise intervention (conventional physical therapy) or a 4-week experimental exercise intervention (plantar flexion training). Both the control and exerimental arms will complete over-ground multi-directional gait training and home exercise.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to perform five times sit to stand test without the use of upper extremities
* Must have 10 degrees of passive ankle dorsiflexion measured in standing
* Must be able to walk with supervision level assistance with no assistive device

Exclusion criteria:

* Currently receiving physical therapy
* History of orthopedic ankle instability
* Lacking knee extension to neutral
* Unable to understand English
* Unable to follow multi-step commands
* History of orthopedic pathology that prevents completion of experimental condition
* Pain with weight bearing on paretic LE
* Received Botox to the plantar flexors within the last three months or phenol injections within the last six months
* Walk with a longer nonparetic step length than paretic step length

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Step length asymmetry ratio as assessed by the GAITRite® | baseline, 6 weeks (relative to the phase 3 intervention)
  The step length asymmetry ratio will be calculated by dividing the paretic step length by non-paretic step lengths. The magnitude of the ratio indicates the nature of the asymmetry, with symmetrical gait defined as step length ratio of 0.9-1.1, and asymmetrical gait where the non-paretic step lengths are longer than the paretic step lengths with any step length ratio greater than 1.1.
Muscle activity of the medial gastrocnemius as assessed by surface EMG | on the 1 day of the phase 1 intervention
  Muscle activity of the medial gastrocnemius will be assessed using surface EMG (Delsys Trigno EMG system, Boston, MA, USA). The EMG instrument will be placed on the muscle belly of medial gastrocnemius muscle in the paretic lower extremity (LE).
Muscle activity of the soleus as assessed by surface EMG | on the 1 day of the phase 1 intervention
  Muscle activity of the medial gastrocnemius will be assessed using surface EMG (Delsys Trigno EMG system, Boston, MA, USA). The EMG instrument will be placed on the muscle belly of soleus muscle in the paretic lower extremity (LE).
Plantar flexion torque as assessed by isokinetic dynamometry | baseline, 6 weeks (relative to the phase 3 intervention)
  Peak plantar flexion torque will be acquired using an isokinetic dynamometer(Biodex Medical Systems, Shirely, New York, USA). Calibration of the Biodex® will be performed prior to the assessment of each individual. For each participant, the plantar flexors will be warmed-up on a LE ergometer for 10 minutes prior to testing. The participant will be fully secured to prevent compensatory behaviors from trunk or hips that may influence results. A pre-speed warm up on the Biodex of three submaximal repetitions and one maximal repetition will be conducted prior to testing so the participant understands what these repetitions feel like. The angular velocity will be set a 60°/second, five repetitions will be performed, and the peak torque of the plantar flexors will be collected.
Muscle activity of the medial gastrocnemius as assessed by surface EMG | on the 1 day of the phase 2 intervention
  Muscle activity of the medial gastrocnemius will be assessed using surface EMG (Delsys Trigno EMG system, Boston, MA, USA). The EMG instrument will be placed on the muscle belly of medial gastrocnemius muscle in the paretic lower extremity (LE).
Muscle activity of the soleus as assessed by surface EMG | on the 1 day of the phase 2 intervention
  Muscle activity of the medial gastrocnemius will be assessed using surface EMG (Delsys Trigno EMG system, Boston, MA, USA). The EMG instrument will be placed on the muscle belly of soleus muscle in the paretic lower extremity (LE).

SECONDARY OUTCOMES:
Gait speed as assessed by the GAITRite® | baseline, 6 weeks (relative to the phase 3 intervention)
  Self-selected gait speed will be acquired using the GAITRite®.
Muscle activity of the medial gastrocnemius as assessed by surface EMG | baseline, 6 weeks (relative to the phase 3 intervention)
  Muscle activity of the medial gastrocnemius will be assessed using surface EMG (Delsys Trigno EMG system, Boston, MA, USA). The EMG instrument will be placed on the muscle belly of medial gastrocnemius muscle in the paretic lower extremity (LE).
Muscle activity of the soleus as assessed by surface EMG | baseline, 6 weeks (relative to the phase 3 intervention)
  Muscle activity of the medial gastrocnemius will be assessed using surface EMG (Delsys Trigno EMG system, Boston, MA, USA). The EMG instrument will be placed on the muscle belly of soleus muscle in the paretic lower extremity (LE).
Quality of life as assessed by the Stroke Impact Scale | baseline, 6 weeks (relative to the phase 3 intervention)
  The physical domain of the Stroke Impact Scale will used to determine quality of life. The Stroke Impact Scale is a self-report measure designed to capture eight domains of health status. The physical domain has nine items that are rated using a 5 point Likert scale in terms of how difficult certain physical tasks are. The domains are scored separately using a transformed scale formula: [(raw score - lowest possible raw score) / highest possible raw score] x 100. A composite score will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P Wingard, DPT, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States